CLINICAL TRIAL: NCT02161679
Title: Randomized Phase II Study of IMMU-132 Alone or in Combination With Carboplatin in Patients With Relapsed/Refractory Triple-Negative Breast Cancer
Brief Title: Phase II Study of IMMU-132 Alone or in Combination With Carboplatin in Patients With Triple-Negative Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA asked to administratively split from IND115621- to open a new IND you need to file a protocol we only drafted it to get the IND open - never initiated
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMMU-132-02
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2020-09

CONDITIONS: Triple-negative Breast Cancer
Keywords: Antibody drug conjugate; IMMU-132; Triple-negative breast cancer; Safety and tolerability; Progression Free Survival (PFS)
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan

ARMS (2):
- IMMU-132 (Experimental): IMMU-132 infusion is administered
  Interventions: Drug: IMMU-132 infusion is administered to participants in one arm for the study; Drug: IMMU-132 plus Carboplatin infusion
- IMMU-132 plus Carboplatin (Active Comparator): IMMU-132 infusion and Carboplatin infusion are administered to the participants in this arm of study.
  Interventions: Drug: IMMU-132 infusion is administered to participants in one arm for the study; Drug: IMMU-132 plus Carboplatin infusion

INTERVENTIONS:
Drug: IMMU-132 infusion is administered to participants in one arm for the study
Drug: IMMU-132 plus Carboplatin infusion
  Other Names: IMMU-132 and Carboplatin infusions are administered to the participants in this arm of study

SUMMARY:
This is a Phase II, open-label study that evaluates the safety and efficacy of IMMU-132 alone and in combination with carboplatin in patients with triple-negative breast cancer. IMMU132 will be administered once-weekly for the first 2 weeks of 3-week treatment cycles. For those patients assigned to also receive carboplatin, will receive it on the same schedules starting 30 minutes after the completion of IMMU-132 administration. Patients may receive up to a maximum total of 8 cycles.

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety and efficacy of IMMU-132 alone and in combination with carboplatin administered in 3-week treatment cycles for up to 8 cycles, in patients with triple-negative breast cancer that have received at least two prior treatments. The secondary objectives are to obtain data concerning pharmacokinetics, and immunogenicity.

This is a multi-center study. Eighty patients are planned to be enrolled, with an equal distribution between the two groups. All patients will receive a starting dose of IMMU-132administered once-weekly for the first 2 weeks of 3-week treatment cycles. For those patients assigned to also receive carboplatin, carboplatin will also be administered on the same schedules starting 30 minutes after the completion of IMMU-132 administration. Patients may receive up to a maximum total of 8 cycles (16 doses), but patients with a complete response, partial response or stable disease at that time, or patients who had achieved an objective response, but relapsed after discontinuing treatment, may continue to be treated based on physician discretion. Follow up is then required until resolution or stabilization of any treatment-related toxicity, and patients with stable disease or objective responses must also continue evaluations until survived.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with triple negative metastatic breast cancer, age 18 years or older, pathologically confirmed metastatic adenocarcinoma of the breast. Pathologically confirmed as triple-negative, measurable disease, defined by (RECIST 1.1) guidelines;
* Two or more prior chemotherapy, immunotherapy and/or monoclonal antibody therapy for the treatment of the subjects' metastatic breast cancer;
* Prior neoadjuvant or adjuvant chemotherapy must have been completed at least 4 weeks before start of study treatment with all related toxicities resolved;
* Prior radiotherapy must have completed at least 2 weeks before randomization, with full recovery;
* At least 4 weeks from major surgery, ECOG performance status 0-1.
* Hematology parameters (ANC) ≥ 1500/mm2;
* Platelets ≥ 100,000/mm2;
* Hemoglobin (Hgb) ≥ 9 g/dL AST & ALT ≤ 2.5 x ULN);
* If hepatic metastases present ≤ 5.0 x ULN Total bilirubin ≤ ULN ;
* Subjects with Gilbert's syndrome can have bilirubin of up to 1.5 x ULN;
* Alkaline phosphatase ≤ 2.5 x ULN (unless bone metastases are present in the absence of liver metastasis);
* Creatinine clearance > 60 mL/min

Exclusion Criteria:

* Male subjects with triple negative metastatic breast cancer;
* Concurrent chemotherapy, immunotherapy or monoclonal antibody or any other anti-tumor therapy for breast cancer,
* Concurrent or prior anticoagulation therapy within 7 days of first dose of study treatment,
* History of, or known current evidence of brain metastasis, including leptomeningeal involvement;
* Subjects with bone as the only site of metastatic disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years